CLINICAL TRIAL: NCT06414837
Title: Study on Efficacy and Safety of HR091506 Tablets in Treatment of Gout With Hyperuricemia in Adults
Brief Title: Clinical Trial of HR091506 Tablets in Treatment of Gout With Hyperuricemia in Adults
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR091506-301
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Gout With Hyperuricemia in Adults
MeSH Terms: interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A: HR091506 tablets + placebo of febuxostat tablets (Experimental)
  Interventions: Drug: HR091506 tablets + placebo of febuxostat tablets
- Treatment group B: febuxostat tablets + placebo of HR091506 tablets (Active Comparator)
  Interventions: Drug: febuxostat tablets + placebo of HR091506 tablets

INTERVENTIONS:
Drug: HR091506 tablets + placebo of febuxostat tablets — HR091506 tablets 20mg/ 40mg/ 60mg/80mg qd + placebo of febuxostat tablets 20mg/ 40mg/ 60mg/80mg qd, from Week 1 to 36.
  Arms: Treatment group A: HR091506 tablets + placebo of febuxostat tablets
Drug: febuxostat tablets + placebo of HR091506 tablets — febuxostat tablets 20mg/ 40mg/ 60mg/80mg qd + placebo of HR091506 tablets 20mg/ 40mg/ 60mg/80mg qd . from Week 1 to 36.
  Arms: Treatment group B: febuxostat tablets + placebo of HR091506 tablets

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of HR091506 tablets for treatment of gout with hyperuricemia in adults, and to compare the results with febuxostat tablets in the same doses.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, male or female;
2. Meet the 2015 ACR/EULAR gout classification criteria;
3. Fast serum uric acid ≥ 480 μmol/L on 2 different days during the screening perid;
4. Patients with tophi, chronic arthropathy, frequent attacks;
5. Willing to ues contraceptive measures during the study;
6. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. History of acute gout attack within 4 weeks before randomization.
2. Subjects who have undergone major surgery or organ transplantation within 3 months before randomization.
3. Subjects with major cardiovascular disease within 6 months before randomization.
4. History of chronic infection or recurrent infection within 1year before randomization.
5. History of malignant tumor or current history of combined malignant tumor within 5 years before screening.
6. History of secondary hyperuricemia, refractory gout, or xanthine metabolism disorder.
7. Subjects with poorly controlled blood pressure or diabetes mellitus.
8. History of chronic diffuse connective tissue disease and/or massively elevated urate diseases and/or untreated clinically significant thyroid disease.
9. History of diseases that may affect the in vivo process, safety evaluation, or subjects' participation in the research.
10. Abnormal laboratory tests that may affect subjects participating in the research.
11. Combined use of prohibited drugs.
12. Allergic to ingredient or component of the experimental drug.
13. Participated in other clinical trials within 1 month before randomization.
14. Pregnant or nursing women.
15. History of drug abuse, drug use and/or excessive drinking within 1 year before screening.
16. The inestigators determined that other conditions were inappropriate for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with serum uric acid level < 300 μmoL/L at Week 36 | Week 36

SECONDARY OUTCOMES:
Proportion of subjects with serum uric acid level < 360 μmol/L at week 4,8,12,16,20,24,28,32,36 after administration | at week 4,8,12,16,20,24,28,32,36 after administration
Proportion of subjects with serum uric acid level < 300 μmol/L at week 4,8,12,16,20,24,28,32,36 after administration | at week 4,8,12,16,20,24,28,32,36 after administration
Change of serum uric acid level from baseline week 4,8,12,16,20,24,28,32,36 after administration | week 4,8,12,16,20,24,28,32,36 after administration
Proportion of subjects with ≥1 gout flare during the 36 weeks treatment stage | during the 36 weeks treatment stage

IPD SHARING:
Plan to Share IPD: Undecided